CLINICAL TRIAL: NCT04458662
Title: Iron and Muscular Damage: FEmale Metabolism and Menstrual Cycle During Exercise
Acronym: IronFEMME
Status: Completed | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, ANA BELEN PEINADO LOZANO, Associate Professor, Universidad Politecnica de Madrid
Other Study IDs: DEP2016-75387-P
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Iron-deficiency; Inflammation; Exercise Induced Iron-deficiency; Exercise Induced Muscle Damage; Regulation of Sex Hormones on Hepcidin; Regulation of Sex Hormones on Muscle Damage; Iron Metabolism Disorders
Keywords: Hepcidin; Iron deficiency; Menstrual cycle; Muscle damage; Creatine kinase; Female; Exercise; Estrogen; Progesterone; Oral contraceptives; Postmenopausal women
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammation; Iron Metabolism Disorders; Iron Deficiencies; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eumenorrheic women: The project consisted on two sections carrying out at the same time: Iron physiology (Study I) and Muscle damage (Study II).
  For the study I, the exercise protocol consisted on an interval running test. 5 min warm-up at 60% of the vVO2peak followed by 8 bouts of 3 min at 85% of the vVO2peak with 90 secs recovery at 30% of the vVO2peak between bouts. Finally, a 5 min cool down was performed at 30% of the vVO2peak.
  The study II protocol was based on an eccentric-based resistance exercise protocol consisted on 10 sets of 10 reps of plate-loaded parallel back squats at 60% of their previously calculated 1RM with 2 mins recoveries between sets.
  In both studies, eumenorrheic participants were evaluated at three specific moments of the menstrual cycle: Early-follicular phase (EFP), late-follicular phase (LFP) and mid-luteal phase (MLP);
  Interventions: Procedure: Interval running protocol / eccentric-based resistance exercise protocol
- Oral contraceptive users: The project consisted on two sections carrying out at the same time: Iron physiology (Study I) and Muscle damage (Study II).
  For the study I, the exercise protocol consisted on an interval running test. 5 min warm-up at 60% of the vVO2peak followed by 8 bouts of 3 min at 85% of the vVO2peak with 90 secs recovery at 30% of the vVO2peak between bouts. Finally, a 5 min cool down was performed at 30% of the vVO2peak.
  The study II protocol was based on an eccentric-based resistance exercise protocol consisted on 10 sets of 10 reps of plate-loaded parallel back squats at 60% of their previously calculated 1RM with 2 mins recoveries between sets.
  Oral contraceptive users performed the trial at two moments: Withdrawal phase (WP) and active pill phase (APP).
  Interventions: Procedure: Interval running protocol / eccentric-based resistance exercise protocol
- Postmenopausal women: he project consisted on two sections carrying out at the same time: Iron physiology (Study I) and Muscle damage (Study II).
  For the study I, the exercise protocol consisted on an interval running test. 5 min warm-up at 60% of the vVO2peak followed by 8 bouts of 3 min at 85% of the vVO2peak with 90 secs recovery at 30% of the vVO2peak between bouts. Finally, a 5 min cool down was performed at 30% of the vVO2peak.
  The study II protocol was based on an eccentric-based resistance exercise protocol consisted on 10 sets of 10 reps of plate-loaded parallel back squats at 60% of their previously calculated 1RM with 2 mins recoveries between sets.
  Postmenopausal women were tested only once, since their hormonal status does not fluctuate.
  Interventions: Procedure: Interval running protocol / eccentric-based resistance exercise protocol

INTERVENTIONS:
Procedure: Interval running protocol / eccentric-based resistance exercise protocol

SUMMARY:
This project is an observational controlled randomized counterbalance study. One hundred and three physically active and healthy women were selected to participate in the IronFEMME Study, of which 57 were eumenorrheic, 30 were oral contraceptive users (OCP) and 16 were postmenopausal women. The project consisted on two sections carrying out at the same time: Iron metabolism (Study I) and Muscle damage (Study II). For the study I, the exercise protocol consisted on an interval running test (8 bouts of 3 min at 85% of the maximal aerobic speed), whereas the study II protocol was based on an eccentric-based resistance exercise protocol (10 sets of 10 repetitions of plate-loaded barbell parallel back squats at 60% of their 1RM with 2 min of rest between sets). In both studies, eumenorrheic participants were evaluated at three specific moments of the menstrual cycle: Early-follicular phase, late-follicular phase and mid-luteal phase; OCP performed the trial at two moments: Withdrawal phase and active pill phase. Lastly, postmenopausal women were tested only once, since their hormonal status does not fluctuate. The three-step method was used to verify the menstrual cycle phase: calendar counting, blood analyses confirmation and urine-based ovulation kits. Blood samples were obtained to measure sexual hormones (e.g., 17β-Estradiol, Progesterone), iron metabolism parameters (e.g., Hepcidin, Iron, Ferritin, Transferrin) and muscle damage related markers (e.g., Creatine Kinase, Myoglobin, Lactate Dehydrogenase).

ELIGIBILITY:
Inclusion Criteria:

Participants were required to meet the following criteria:

* Healthy adult females between 18 and 40 years old for eumerroheic and oral contraceptive groups or under 60 years old for postmenopausal women.
* Presenting with healthy iron parameters (serum ferritin >20μg/l, haemoglobin >115 μg/l and transferrin saturation >16%).
* Performing endurance training between 5 and 12 h per week (study I) or experienced in resistance training performing at least 1 h session two times per week during a minimum of a year (study II).

Exclusion Criteria:

The exclusion criteria included:

* Irregular menstrual cycles.
* Any existing disease and/or metabolic or hormonal disorder.
* Any musculoskeletal injury in the last six months prior to the beginning of the project.
* Any surgery interventions (e.g. ovariectomy) or other medical conditions that would be exacerbated by an eccentric resistance exercise protocol.
* Regular use of medication or dietary supplements that could affect the results (e.g. nonsteroidal anti-inflammatory drugs).
* Taking medication that alters vascular function (e.g. tricyclic antidepressants, α-blockers, β-blockers, etc.).
* Pregnancies in the year preceding.
* Smoking.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physically active and healthy women. Study I, 37 eumenorrheic women (30.0±6.3 yrs; 59.8±15.7 kg; 163.7±6.3 cm): endurance training (ET) experience of 7.7 yrs and training volume of 5.5±0.9 h/week. Study II, 20 eumenorrheic women (28.8±6.2 yrs; 57.5±13.8 kg; 163.9±6.4 cm): strength training (ST) experience of 6.4±4.1 yrs and training volume of 7.5±2.1 h/week. Eumenorrheic women selected to participate in Study I and II were different, whereas oral contraceptive users and postmenopausal women participated in both studies. 30 oral contraceptive users (25.1±4.3 yrs; 56.2±10.9 kg; 163.1±5.5 cm): ET experience of 7.3±5.5 yrs and training volume of 3.4±1.5 h/week; ST experience of 3.1±1.9 yrs and training volume of 2.5±1.4 h/week. 16 postmenopausal women (51.4±3.7 yrs; 56.7±8.3 kg; 161.7±4.9 cm): ET experience of 7.9±3.4 yrs and training volume of 4.1±1.2 h/week; ST experience of 3.1±1.9 yrs and training volume of 1.6±0.9 h/week
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Hepcidin | pre-exercise
  Hepcidin is a protein that in humans is encoded by the HAMP gene. Hepcidin is a key regulator of the entry of iron into the circulation in mammals
Hepcidin | 0 hours post-exercise
  Hepcidin is a protein that in humans is encoded by the HAMP gene. Hepcidin is a key regulator of the entry of iron into the circulation in mammals
Hepcidin | 3 hours post-exercise
  Hepcidin is a protein that in humans is encoded by the HAMP gene. Hepcidin is a key regulator of the entry of iron into the circulation in mammals
Hepcidin | 24 hours post-exercise
  Hepcidin is a protein that in humans is encoded by the HAMP gene. Hepcidin is a key regulator of the entry of iron into the circulation in mammals
Creatine kinase | pre-exercise
  It is an enzyme that helps regulate the concentration of adenosine triphosphate within a cell. To do so, creatine kinase catalyzes the movement of a phosphate group from ATP to creatine, forming phosphocreatine. This molecules stores the phosphate group in a stable form, acting as an energy reservoir in cells.
Creatine kinase | 2 hours post-exercise
  It is an enzyme that helps regulate the concentration of adenosine triphosphate within a cell. To do so, creatine kinase catalyzes the movement of a phosphate group from ATP to creatine, forming phosphocreatine. This molecules stores the phosphate group in a stable form, acting as an energy reservoir in cells.
Creatine kinase | 24 hours post-exercise
  It is an enzyme that helps regulate the concentration of adenosine triphosphate within a cell. To do so, creatine kinase catalyzes the movement of a phosphate group from ATP to creatine, forming phosphocreatine. This molecules stores the phosphate group in a stable form, acting as an energy reservoir in cells.
Creatine kinase | 48 hours post-exercise
  It is an enzyme that helps regulate the concentration of adenosine triphosphate within a cell. To do so, creatine kinase catalyzes the movement of a phosphate group from ATP to creatine, forming phosphocreatine. This molecules stores the phosphate group in a stable form, acting as an energy reservoir in cells.

SECONDARY OUTCOMES:
Iron | pre-exercise
Iron | 0 hours post-exercise
Iron | 3 hours post-exercise
Iron | 24 hours post-exercise
Transferrin | pre-exercise
Transferrin | 0 hours post-exercise
Transferrin | 3 hours post-exercise
Transferrin | 24 hours post-exercise
Ferritin | pre-exercise
Ferritin | 0 hours post-exercise
Ferritin | 3 hours post-exercise
Ferritin | 24 hours post-exercise
Mioglobin | pre-exercise
Mioglobin | 2 hours post-exercise
Mioglobin | 24 hours post-exercise
Mioglobin | 48 hours post-exercise
LDH | pre-exercise
  Lactate deshidrogenase
LDH | 2 hours post-exercise
  Lactate deshidrogenase
LDH | 24 hours post-exercise
  Lactate deshidrogenase
LDH | 48 hours post-exercise
  Lactate deshidrogenase
TNF-alfa | pre-exercise
TNF-alfa | 2 hours post-exercise
TNF-alfa | 24 hours post-exercise
TNF-alfa | 48 hours post-exercise
Interleukin-6 | pre-exercise
Interleukin-6 | 0 hours post-exercise
Interleukin-6 | 2 hours post-exercise
Interleukin-6 | 24 hours post-exercise
Interleukin-6 | 48 hours post-exercise
CRP | pre-exercise
  C-reactive protein
CRP | 0 hours post-exercise
  C-reactive protein
CRP | 2 hours post-exercise
  C-reactive protein
CRP | 24 hours post-exercise
  C-reactive protein
CRP | 48 hours post-exercise
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Ana Belén Peinado, Study Director — LFE Research Group. Universidad Politécnica de Madrid
Locations (1):
- Laboratorio de Fisiología Del Esfuerzo. Facultad de Ciencias de La Actividad Física Y Del Deporte. Universidad Politécnica de Madrid., Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehtihet M, Bonde Y, Beckman L, Berinder K, Hoybye C, Rudling M, Sloan JH, Konrad RJ, Angelin B. Circulating Hepcidin-25 Is Reduced by Endogenous Estrogen in Humans. PLoS One. 2016 Feb 11;11(2):e0148802. doi: 10.1371/journal.pone.0148802. eCollection 2016. PMID 26866603
- [Background] Hou Y, Zhang S, Wang L, Li J, Qu G, He J, Rong H, Ji H, Liu S. Estrogen regulates iron homeostasis through governing hepatic hepcidin expression via an estrogen response element. Gene. 2012 Dec 15;511(2):398-403. doi: 10.1016/j.gene.2012.09.060. Epub 2012 Oct 3. PMID 23041085
- [Background] Ikeda Y, Tajima S, Izawa-Ishizawa Y, Kihira Y, Ishizawa K, Tomita S, Tsuchiya K, Tamaki T. Estrogen regulates hepcidin expression via GPR30-BMP6-dependent signaling in hepatocytes. PLoS One. 2012;7(7):e40465. doi: 10.1371/journal.pone.0040465. Epub 2012 Jul 11. PMID 22792339
- [Background] Li X, Rhee DK, Malhotra R, Mayeur C, Hurst LA, Ager E, Shelton G, Kramer Y, McCulloh D, Keefe D, Bloch KD, Bloch DB, Peterson RT. Progesterone receptor membrane component-1 regulates hepcidin biosynthesis. J Clin Invest. 2016 Jan;126(1):389-401. doi: 10.1172/JCI83831. Epub 2015 Dec 14. PMID 26657863
- [Background] Yang Q, Jian J, Katz S, Abramson SB, Huang X. 17beta-Estradiol inhibits iron hormone hepcidin through an estrogen responsive element half-site. Endocrinology. 2012 Jul;153(7):3170-8. doi: 10.1210/en.2011-2045. Epub 2012 Apr 25. PMID 22535765
- [Background] Thompson B, Almarjawi A, Sculley D, Janse de Jonge X. The Effect of the Menstrual Cycle and Oral Contraceptives on Acute Responses and Chronic Adaptations to Resistance Training: A Systematic Review of the Literature. Sports Med. 2020 Jan;50(1):171-185. doi: 10.1007/s40279-019-01219-1. PMID 31677121
- [Background] McClung JP. Iron status and the female athlete. J Trace Elem Med Biol. 2012 Jun;26(2-3):124-6. doi: 10.1016/j.jtemb.2012.03.006. Epub 2012 May 7. PMID 22572041
- [Background] Kendall B, Eston R. Exercise-induced muscle damage and the potential protective role of estrogen. Sports Med. 2002;32(2):103-23. doi: 10.2165/00007256-200232020-00003. PMID 11817996
- [Background] Tiidus PM, Lowe DA, Brown M. Estrogen replacement and skeletal muscle: mechanisms and population health. J Appl Physiol (1985). 2013 Sep 1;115(5):569-78. doi: 10.1152/japplphysiol.00629.2013. Epub 2013 Jul 18. PMID 23869062
- [Background] Sim M, Dawson B, Landers G, Swinkels DW, Tjalsma H, Yeap BB, Trinder D, Peeling P. Oral contraception does not alter typical post-exercise interleukin-6 and hepcidin levels in females. J Sci Med Sport. 2015 Jan;18(1):8-12. doi: 10.1016/j.jsams.2013.11.008. Epub 2013 Nov 28. PMID 24373771
- [Background] Sipaviciene S, Daniuseviciute L, Kliziene I, Kamandulis S, Skurvydas A. Effects of estrogen fluctuation during the menstrual cycle on the response to stretch-shortening exercise in females. Biomed Res Int. 2013;2013:243572. doi: 10.1155/2013/243572. Epub 2013 Sep 12. PMID 24151587
- [Background] Janse DE Jonge X, Thompson B, Han A. Methodological Recommendations for Menstrual Cycle Research in Sports and Exercise. Med Sci Sports Exerc. 2019 Dec;51(12):2610-2617. doi: 10.1249/MSS.0000000000002073. PMID 31246715
- [Result] Romero-Parra N, Barba-Moreno L, Rael B, Alfaro-Magallanes VM, Cupeiro R, Diaz AE, Calderon FJ, Peinado AB. Influence of the Menstrual Cycle on Blood Markers of Muscle Damage and Inflammation Following Eccentric Exercise. Int J Environ Res Public Health. 2020 Mar 2;17(5):1618. doi: 10.3390/ijerph17051618. PMID 32131554
- [Derived] Guisado-Cuadrado I, Romero-Parra N, Cupeiro R, Elliott-Sale KJ, Sale C, Peinado AB. Effect of eccentric-based resistance exercise on bone (re)modelling markers across the menstrual cycle and oral contraceptive cycle. Eur J Appl Physiol. 2025 May;125(5):1463-1473. doi: 10.1007/s00421-024-05693-y. Epub 2024 Dec 30. PMID 39738864
- [Derived] Guisado-Cuadrado I, Alfaro-Magallanes VM, Romero-Parra N, Rael B, Guadalupe-Grau A, Peinado AB. Influence of sex hormones status and type of training on regional bone mineral density in exercising females. Eur J Sport Sci. 2023 Nov;23(11):2139-2147. doi: 10.1080/17461391.2023.2211947. Epub 2023 May 17. PMID 37161678
- [Derived] Alfaro-Magallanes VM, Barba-Moreno L, Romero-Parra N, Rael B, Benito PJ, Swinkels DW, Laarakkers CM, Diaz AE, Peinado AB; IronFEMME Study Group. Menstrual cycle affects iron homeostasis and hepcidin following interval running exercise in endurance-trained women. Eur J Appl Physiol. 2022 Dec;122(12):2683-2694. doi: 10.1007/s00421-022-05048-5. Epub 2022 Sep 21. PMID 36129579
- See also: IronFEMME project official web page — https://ironfemme.com